CLINICAL TRIAL: NCT04270981
Title: An Open Label, Single-dose, Single Period Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C-Acoziborole
Brief Title: ADME Study of Acoziborole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-OXA-03-HAT
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Trypanosomiases, African
MeSH Terms: conditions — Trypanosomiasis, African

STUDY DESIGN:
Intervention Model Description: single centre, open-label, single group, non-randomised, single oral dose study in healthy male subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-acoziborole capsule, 240 mg containing NMT 9.25 kBq (250 (Experimental): single administration of 960 mg (4 × 240 mg capsules) acoziborole in oral and fasted condition
  Interventions: Drug: [14C]-acoziborole capsule, 240 mg containing NMT 9.25 kBq (250 nCi) 14C

INTERVENTIONS:
Drug: [14C]-acoziborole capsule, 240 mg containing NMT 9.25 kBq (250 nCi) 14C — 960 mg (4 × 240 mg capsules)of acoziborole in oral and fasted condition
  Other Names: no other name

SUMMARY:
This is a single centre, open-label, single group, non-randomised, single oral dose study in healthy male subjects designed to assess the mass balance recovery, PK, metabolite profile and metabolite identification, and exploratory pharmacodynamics of acoziborole. It is planned to enrol 6 subjects.

All subjects will receive an oral dose of 960 mg [14C] acoziborole on a single occasion as 4 capsules containing a small amount of radioactivity (not more than [NMT] 1000 nCi [37 KBq] 14C).

DETAILED DESCRIPTION:
The present study aims to further understand and quantify the absorption, distribution, metabolism and elimination (ADME) of acoziborole in humans through the assessment of the mass balance recovery after a single oral dose of [14C]-acoziborole. The routes and rates of elimination of [14C]-acoziborole will be determined and plasma, urine and faecal samples will be used for metabolic profiling and structural identification.

Subjects will be screened for inclusion in the study up to 28 days before dosing. Subjects will be admitted in the evening on the day before dosing (Day 1).

Subjects will be dosed on the morning of Day 1 following an overnight fast of a minimum of 9 h, and will remain resident in the clinic until up to 240 h after dosing (up to Day 11). Subjects will return to the clinical unit for 5 additional 48 h collection periods, admitting to the clinical unit the evening before the collection period. The additional collection periods will be on Days 14 to 17, 28 to 31, 58 to 61, 88 to 91 and 118 to 121. A follow up call will take place 5 to 10 days post-final discharge to ensure the ongoing wellbeing of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males.
* Age 18 to 55 years of age at the time of signing informed consent.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening.
* Must be willing and able to communicate and participate in the whole study.
* Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day).
* Normal blood pressure (BP): Systolic BP between 90 and 140 (160 if >45 years old) mmHg (inclusive), diastolic BP 45 to 90 mmHg (inclusive), measured after 10 min rest in supine position at screening and pre-dose.
* A resting heart rate (HR) between 45 and 100 bpm (inclusive), measured after 10 min rest in supine position at screening and pre-dose.
* ECG recording without clinically significant abnormality, including QTcF measure of ≤450 msec at screening and pre-dose.
* Must provide written informed consent.
* Must agree to adhere to the contraception requirements
* Subjects must be able to swallow multiple capsules.

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week and (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type) as confirmed by a positive alcohol breath test at screening or any on admission to the clinical unit.
* Current smokers and those who have smoked within the last 6 months. As confirmed by a breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Subjects with pregnant or lactating partners.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 year. No occupationally exposed worker shall participate in the study.
* Subjects who have been enrolled in an ADME study in the last 12 months.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
* Clinically significant abnormal clinical chemistry, haematology, urinalysis (especially alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase) or clinically significant abnormal physical examination findings as judged by the investigator .
* Abnormal thyroid function test results
* Abnormal renal function (estimate glomerular filtration rate [eGFR] <80 mL/min).
* Confirmed positive drugs of abuse test result .
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
* History of any clinically significant acute or chronic cardiovascular, renal, hepatic, neurological (especially seizures), immunological, psychiatric, myopathies, bleeding tendency, respiratory and particularly GI disease, especially peptic ulceration and chronic gastritis, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome, as judged by the investigator.
* Any relevant GI complaints within 7 days of dosing.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment (including asthma, urticaria, clinically significant allergic rash or other severe allergic diathesis), as judged by the investigator. Hay fever is allowed unless it is active.
* Donation or loss of greater than 400 mL of blood within the previous 3 months or more than 100 mL within 30 days before signing ICF to this trial.
* Subjects who are taking any prescribed drug in the 14 days before screening or require regular use of any prescription medication during the study
* Subjects who have taken, any over-the-counter medications, including vitamins, analgesics or antacids, herbal remedies or St. John's wort in the 7 days before IMP administration . Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the PI.
* Use of enzyme-altering drugs (e.g. barbiturates, phenothiazines, cimetidine) within 30 days or 5 half-lives, whichever is longer, of study Day 1.
* Surgery within 12 weeks prior to screening, with the exception of appendectomy or at the discretion of the Investigator for minor surgery.
* Any surgery (e.g. gastric bypass) or medical condition that may affect absorption of orally administered drugs.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
total radioactivity in urines and feces | 121 days
  Total radioactivity in urine and faeces at each time interval and cumulative radioactivity excretion (mass balance). For the sample collection periods following 240 h after the dose, excretion will be interpolated between collection periods

SECONDARY OUTCOMES:
Plasma and urine concentrations of acoziborole and of its main metabolite, SCYX 3109 | 121 days
  Plasma and urine concentrations of acoziborole and of its main metabolite, SCYX 3109, to determine relevant PK parameters
Total radioactivity in whole blood (optional), plasma, urine and faeces | 121 days
  Total radioactivity in whole blood (optional), plasma, urine and faeces at each time point, to determine relevant PK parameters
Quantitative metabolite profiling and identification of metabolites in pooled samples of plasma, urine and faeces | 121 days
  Quantitative metabolite profiling and identification of metabolites in pooled samples of plasma, urine and faeces, using liquid chromatography (LC)/accelerator mass spectrometry (AMS) in conjunction with LC/tandem mass spectrometry (MS-MS)
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with adverse events | 126 days
  Safety and tolerability of 14C acoziborole after single dose as measured by d number of subjects with adverse events
safety and tolerability of 14C acoziborole after single dose as measured by adverse events severity | 126 days
  Safety and tolerability of 14C acoziborole after single dose as measured by adverse events severity
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with vital signs findings | 121 days
  Safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with vital signs findings
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with 12 -lead ECG findings | 121 days
  Safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with 12 -lead ECG findings
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with clinical laboratory tests findings (hematology) | 121 days
  Safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with clinical laboratory tests findings (hematology)
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with clinical laboratory tests findings (biochemistry) | 121 days
  Safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with clinical laboratory tests findings (biochemistry)
safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with physical examination findings | 121 days
  Safety and tolerability of 14C acoziborole after single dose as measured by number of subjects with physical examination findings
Amount of radioactivity in plasma, faeces and urine over time | 121 days
  Amount of radioactivity in plasma, faeces and urine over time exploratory and optional

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No